CLINICAL TRIAL: NCT05035043
Title: The Economic Burden of Non-Alcoholic Fatty Liver Disease Patients in Flanders, Belgium
Brief Title: Economic Burden of NAFLD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasselt University (Other)
Responsible Party: Principal Investigator, Geert Robaeys, Principal Investigator, Hasselt University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: EB-NAFLD-DGP-001
Record Dates: First submitted 2021-08-30; First posted 2021-09-05 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Non-Alcoholic Fatty Liver Disease; NAFLD
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NAFLD patients (Experimental): Non-Alcoholic Fatty Liver Disease patients
  Interventions: Other: Determination of the economic burden NAFLD patients

INTERVENTIONS:
Other: Determination of the economic burden NAFLD patients — Determination of the economic burden NAFLD patients (Healthcare costs, patient costs, burden of disease

SUMMARY:
To determine the economic burden of NAFLD (Non-Alcoholic-Fatty-Liver Disease) patients in Belgium, Flanders by means of a bottom-up approach.

ELIGIBILITY:
Inclusion Criteria:

* having NAFLD as was diagnosed by FibroScan®,
* 18 years or older
* BMI ≥ 25 kg/m²

Exclusion Criteria:

* unable to give informed consent
* >70 years

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
iMTA MCQ | baseline
  Healthcare cost measured with the iMTA MCQ (Institute for Medical Technology Assessment Medical Consumption Questionnaire). The volumes of used healthcare costs were multiplied with the unit costs of these corresponding services.

SECONDARY OUTCOMES:
iMTA MCQ | Baseline
  Patient cost measured with the iMTA MCQ (Institute for Medical Technology Assessment Medical Consumption Questionnaire). The volumes of used healthcare costs were multiplied with the unit costs of these corresponding services.
EuroQol-5D-5L | baseline
  : Health related quality of life questionnaire EuroQol-5D-5L is used. Five levels are score in 5 dimensions. It is scaled from 0 to 100%. A higher score indicates a higher quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Geert Robaeys, prof. dr., Principal Investigator — Hasselt University; Leen Heyens, Study Chair — Hasselt University
Locations (1):
- Hasselt University, Hasselt, Belgium